CLINICAL TRIAL: NCT06184529
Title: VR Regulators: Teaching Adults to Manage Children's Big Emotions Through a Brief Virtual Reality Simulation
Brief Title: Virtual Reality (VR) Regulators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: The Children's Trust, Miami FL (Other)
Responsible Party: Principal Investigator, Jason Jent, Associate Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20231355
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Emotion Regulation
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality Group (Experimental): Participants in this group will receive the virtual reality simulation for up to 6 weeks.
  Interventions: Behavioral: Virtual Reality

INTERVENTIONS:
Behavioral: Virtual Reality — The virtual reality simulation includes a one time viewing of a brief video tutorial and then trying out a one time virtual reality simulation with a child avatar that takes 10-20 minutes to complete in-person.

SUMMARY:
The purpose of this study is to test how well a virtual reality simulation helps adults learn new skills for managing children's emotions.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years old or higher AND
* Caregiver of a child ages 3-6 years old OR educator or child allied health or medical professional that regularly works with children ages 3-6 years old

Exclusion Criteria:

* adults who do not speak English or Spanish
* adults with a history of significant motion sickness, active nausea, and vomiting or epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Adult Emotion Regulation as measured by the Difficulties in Emotion Regulation Scale | Baseline
  Score ranges from 18-90 with higher scores representing more problems with emotion regulation.
Changes in adult responses to child emotions as measured by the Adult Responses to Young Children's Strong Emotions Scale | Baseline, up to 10 minutes post-intervention, 1 month post-intervention
  Score ranges from 7-35 with higher scores representing a higher frequency of reported or planned use of adaptive emotion regulation responses to children

SECONDARY OUTCOMES:
Satisfaction as measured by the Virtual Reality Satisfaction Survey | up to 10 minutes post-intervention
  Score ranges from 5-25 with higher scores representing higher satisfaction with the virtual reality simulation

CONTACTS AND LOCATIONS:
Overall Officials: Jason Jent, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No